CLINICAL TRIAL: NCT07377968
Title: Efficacy of Wearable Device to Promote CPAP Adherence in Patients With Obstructive Sleep Apnea (OSA); A Randomized Controlled Trial
Brief Title: Wearable Device to Promote CPAP Adherence in Obstructive Sleep Apnea (OSA) Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Visasiri Tantrakul, Principal investigator, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: COA. No. MURA2025/1065
Record Dates: First submitted 2026-01-05; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: adherence; OSA; wearable device; health
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wearable group (Experimental): Standard care of CPAP with Garmin vivoactive 5 with self-monitoring data (Patients can access the data by themselves)
  Interventions: Device: garmin vivoactive 5 with self-monitoring data
- Control group (Sham Comparator): Standard care of CPAP with Garmin vivoactive 5 no self-monitoring data (Patients cannot access the data by themselves)
  Interventions: Device: Garmin vivoactive 5 without self-monitoring data

INTERVENTIONS:
Device: garmin vivoactive 5 with self-monitoring data — patients can access health data by themselves
  Arms: Wearable group
Device: Garmin vivoactive 5 without self-monitoring data — Patients cannot access their health data
  Arms: Control group

SUMMARY:
The goal of this study type: clinical trial is to evaluate adherence for CPAP used with wearable device in OSA patients comparing with controlled group; could include any of the following: adult patients (≥ 19 yr of age) with moderate to severe OSA (AHI ≥ 15 events/hr by polysomnography (PSG), according to the American Academy of Sleep Medicine, diagnosed at the sleep clinic in Ramathibodi hospital, patients with OSA who are first time to prescribed CPAP treatment and in the waiting process for their machine. The main question it aims to answer is: Could a wearable device help increase the adherence of CPAP in obstructive sleep apnea patients?

Primary outcome is adherence for CPAP: time usage per day(min) and % usage > 4 hours

Secondary outcome are access sleepiness and quality of sleep by questionnaire (ESS and PSQI) in Thai version, the correlation between wearable-derived and CPAP data: Total sleep time(min), sleep stage (light, deep and REM), and health information: heart rate, oxygen saturation, stress, sleep score and step counting

If there is a comparison group: Researchers will compare wearable group and control group to see the effect of wearable to increase adherence of CPAP used.

Participants will

* Divide into two group by randomization using 4 block randomization
* In wearable group, the participants will receive wearable and download application, they allow to access all the time
* In control group, the participants will receive wearable and download application, but they will not allow to access until they come to hospital for follow up at the end of the study

DETAILED DESCRIPTION:
1. Lead-in Period Patients who have been diagnosed with moderate to severe obstructive sleep apnea and are scheduled to receive continuous positive airway pressure (CPAP) therapy will be referred to the Sleep Clinic, 7th Floor, Phra Thep Building, Ramathibodi Hospital. At this clinic, the research team will provide detailed information about the study. If the patient agrees to participate, written informed consent will be obtained. Participants will then be randomly assigned into one of two groups - the wearable device group or the control group - using block randomization. The allocation sequence will be prepared by a statistician and sealed in opaque envelopes to maintain allocation concealment. During this period, while waiting for CPAP device delivery from the supplier, participants will be asked to wear a Garmin Vivoactive 5 smartwatch to collect baseline data. They will also complete standardized questionnaires in Thai: the Epworth Sleepiness Scale (ESS) and the Pittsburgh Sleep Quality Index (PSQI) to evaluate baseline sleepiness and sleep quality.
2. Wearable Device Group (N = 40) Participants in this group will receive a Garmin Vivoactive 5 smartwatch and be instructed on its proper use. They will also learn how to access their health data via the Garmin Connect application, including sleep stages (light, deep, REM), heart rate, oxygen saturation, and daily step count. These data will be used to enhance patient engagement and support goal setting for personal health improvement. Participants will continue to receive standard education and counseling regarding CPAP use, with an emphasis on adherence and motivation to achieve optimal health outcomes.
3. Control Group (N = 40) Participants in this group will also receive a Garmin Vivoactive 5 smartwatch but will be informed that access to health data through the application will only be available during follow-up visits at the hospital, including the final follow-up visit. Participants will not have direct access to the application, as login requires a password controlled by the research team. If a participant connects the device to another account, the research team will be able to detect it due to the creation of a new user profile, resulting in incomplete data continuity. Patients will be able to view limited on-screen information, such as average oxygen saturation, sleep score, and step count. The screen brightness will be adjusted to the lowest level to minimize light exposure during sleep. They will also receive standard CPAP education identical to the intervention group, encouraging consistent device use for optimal treatment benefits.
4. Follow-Up Procedures 4.1 Week 1 and 2 (Line call/video call Follow-Up) All participants will be contacted by Line call/video call at Week 1 and 2 to assess CPAP adherence, address difficulties, and provide additional guidance to promote usage of at least 4 hours per night. Participants in the wearable group will be asked to capture screenshots from their Garmin Connect app and send them via the Sleep Center's official LINE account. The data collected will include sleep stage distribution, total sleep time, heart rate, oxygen saturation, sleep score, and step count.

   4.2 Weeks 4 and 8 (Clinic Follow-Up) At Weeks 4 and 8, participants will attend in-person follow-up visits at the Sleep Clinic.

   Data collected will include:
   * From Garmin Connect: sleep stage, total sleep time, HR, oxygen saturation, sleep score, step count.
   * From CPAP device downloads: average usage time per day (minutes), % nights used >4h, AHI, leak, and pressure levels. At Week 8, participants will again complete ESS and PSQI (Thai versions) to evaluate post-intervention outcomes.
5. Data Management and API Integration During the study, the research team will request access to Garmin Health API for raw data retrieval, which may be used for further research analysis or development of a web-based application for patient monitoring.
6. Data Collection and Analysis All collected data will be compiled, cleaned, and analyzed according to the predefined statistical plan.
7. End of Study Procedure At the end of the 8-week study period, participants will return the Garmin Vivoactive 5 smartwatch. The research team will verify data completeness, clean and reset the devices, and prepare them for use by subsequent participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 19 yr of age) with moderate to severe OSA (AHI ≥ 15 events/hr at the sleep clinic in Ramathibodi hospital
* Study after EC approval to March, 2026
* Patients with OSA who are prescribed CPAP therapy and accepted a trial of therapy

Exclusion Criteria:

* Patients deny to provide an informed consent
* Patients had active cardiovascular, pulmonary, psychiatric disease, and epilepsy
* Patients had been previously used CPAP for treatment of OSA
* Patients have a problem to use a wearable device or watch
* Patients had used any smartwatch before
* Patients do not have a smart phone

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-06 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Average daily CPAP usage time | From enrollment to 4 weeks and 8 weeks of treatment
  Average CPAP usage time per day, measured in minutes using CPAP device data.
Percentage of nights with CPAP usage ≥ 4 hours | From enrollment to 4 weeks and 8 weeks of treatment
  Percentage of days with CPAP usage ≥ 4 hours per night, reported as a percentage (%), derived from CPAP device data.

SECONDARY OUTCOMES:
Daytime sleepiness assessed by Epworth Sleepiness Scale (Thai version) | From enrollment to 4 week and 8 week of treament
  Epworth Sleepiness Scale (ESS) total score ranging from 0 to 24; higher scores indicate greater daytime sleepiness. A score >10 indicates excessive daytime sleepiness.
Sleep quality assessed by Pittsburgh Sleep Quality Index (Thai version) | From enrollment to 4 week and 8 week of treatment
  Pittsburgh Sleep Quality Index (PSQI) total score ranging from 0 to 21; higher scores indicate poorer sleep quality. A score >5 indicates poor sleep quality.
Total sleep time | From enrollment to 4 week and 8 week of treatment
  Total sleep time measured in minutes, derived from Garmin Vivoactive 5 and CPAP data
Percentage of light sleep stage derived from wearable device | From enrollment to 4 weeks and 8 weeks of treatment
  Percentage of light sleep stage (%), derived from Garmin Vivoactive 5.
Percentage of deep sleep stage derived from wearable device | From enrollment to 4 weeks and 8 weeks of treatment
  Percentage of deep sleep stage (%), derived from Garmin Vivoactive 5.
Percentage of REM sleep stage derived from wearable device | From enrollment to 4 weeks and 8 weeks of treatment
  Percentage of REM sleep stage (%), derived from Garmin Vivoactive 5.
Mean heart rate derived from wearable device | From enrollment to 4 weeks and 8 weeks of treatment
  Average heart rate measured in beats per minute (bpm), derived from Garmin Vivoactive 5.
Average oxygen saturation derived from wearable device | From enrollment to 4 weeks and 8 weeks of treatment
  Average oxygen saturation measured as a percentage (%), derived from Garmin Vivoactive 5.
Stress score derived from wearable device | From enrollment to 4 weeks and 8 weeks of treatment
  Stress score reported by Garmin Vivoactive 5, ranging from 0 to 100.
Sleep score derived from wearable device | From enrollment to 4 weeks and 8 weeks of treatment
  Sleep score reported by Garmin Vivoactive 5, ranging from 0 to 100.
Daily step count derived from wearable device | From enrollment to 4 weeks and 8 weeks of treatment
  Average daily step count measured in steps per day, derived from Garmin Vivoactive 5.

CONTACTS AND LOCATIONS:
Overall Officials: Visasiri Tantrakul, Doctor of Medicine (M.D.), Principal Investigator — Ramathibodi hospital, Mahidol university
Locations (1):
- Ramathibodi hospital, Mahidol university, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Quintana RP, Lasslo A, Queen GS. Surface activity and human blood platelet aggregation-inhibitory potency. Chem Biol Interact. 1982 Jan;38(2):135-44. doi: 10.1016/0009-2797(82)90035-7. PMID 7055847
- [Background] Moscovice IS. Rural hospitals: a literature synthesis and health services research agenda. Health Serv Res. 1989 Feb;23(6):891-930. PMID 2645251
- [Background] Park GS, Miller EJ Jr. Surgical treatment of stress urinary incontinence: a comparison of the Kelly plication, Marshall-Marchetti-Krantz, and Pereyra procedures. Obstet Gynecol. 1988 Apr;71(4):575-9. PMID 3353049
- [Background] Massachusetts. Supreme Judicial Court. Baird v. Attorney General. 25 Jan 1977. North East Rep Second Ser. 1977;360:288-303. No abstract available. PMID 12038347
- [Background] Sato K, Sato F. Nonisotonicity of simian eccrine primary sweat induced in vitro. Am J Physiol. 1987 Jun;252(6 Pt 2):R1099-105. doi: 10.1152/ajpregu.1987.252.6.R1099. PMID 3296789

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT07377968/Prot_SAP_000.pdf